CLINICAL TRIAL: NCT00926445
Title: Effect of Neonatal Pain- and Distress Experiences on Later Pain Behaviour of Former Preterm and Critically Ill Newborn Infants
Brief Title: Neonatal Pain- and Distress Experiences and Later Pain Behavior of Former Preterm and Critically Ill Newborn Infants
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Cologne (Other)
Responsible Party: University of Cologne, Christoph Huenseler
Other Study IDs: 08-177
Record Dates: First submitted 2009-06-22; First posted 2009-06-23 (Estimated); Last update posted 2009-06-23 (Estimated); Status verified 2009-06

CONDITIONS: Pain
Keywords: Pain behavior
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Saliva for measuring cortisol levels
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Preterm (BW < 1500 grams)
- Critically ill term newborn: ventilation > 48 hours
- Healthy term newborn

SUMMARY:
Preterm and critically ill neonates experience many painful manipulations. The aim of the study is to evaluate the influence of these experiences and maternal deprivation on later pain behavior. Using Scoring systems, Prechtl general movements, skin conductance, testing flexor reflex levels with von Frey filaments and measuring salivary cortisol levels the investigators compare pain behavior of preterm (birth weight (BW) < 1500 grams), term neonates with need of ventilation (> 48 hours) with healthy neonates at the time of their first vaccination at the age of 3-4 months. The investigators are also testing flexor reflexes and skin conductance and general movements in regular intervals during the initial hospital stay. The investigators hypothesize that pain behavior is different at the age of 3-4 months in children with many early painful experiences.

ELIGIBILITY:
Inclusion Criteria:

* Preterm < 1500 grams BW, critically ill term newborn on ventilation > 48 hours

Exclusion Criteria:

* Asphyxia
* ICH grade 3 and higher

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature, critically ill term infants are recruited from the NICU of the University hospital of Cologne. Healthy newborns are recruited from the nursery of the University hospital of Cologne.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2008-11

CONTACTS AND LOCATIONS:
Locations (1):
- Neonatologische Intensivstation, Cologne, North Rhine-Westphalia, Germany